CLINICAL TRIAL: NCT06382532
Title: Biological Diagnostic Techniques for the Diagnosis of Depressive Disorders Malinger Based on the Niacin Skin Response Test (NSRT)
Brief Title: Diagnosis of Depressive Disorder Malinger Using the Niacin Skin Response Test (NSRT)
Status: Not yet recruiting | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Jin Wang, Principal Investigator, Air Force Military Medical University, China
Other Study IDs: AFMMUChina_NSRT
Record Dates: First submitted 2024-04-17; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Depressive Disorder; Malingering
MeSH Terms: conditions — Depressive Disorder; Malingering

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control group: 1. M.I.N.I scale rating without any mental disorder;
  2. Patient Health Questionnaire (PHQ-9) < 5;
  3. No history of mental illness, no family genetic history;
  4. Age 18-60 years old, Males;
  5. Voluntary informed consent form.
  Interventions: Diagnostic Test: Niacin skin reaction test
- Depressive disorder group: 1. Patients with a first depressive disorder meeting DSM-5 criteria;
  2. Age 18-60 years, Males;
  3. Voluntary informed consent.
  Interventions: Diagnostic Test: Niacin skin reaction test
- Depressive disorder malinger group: 1. Clinical complaints meeting Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for the diagnosis of depressive disorder;
  2. Patients with first-episode fraudulent disease who meet the DSM-5 criteria for the diagnosis of Z76.5;
  3. Age 18-60 years, Males;
  4. Voluntary informed consent.
  Interventions: Diagnostic Test: Niacin skin reaction test

INTERVENTIONS:
Diagnostic Test: Niacin skin reaction test — Nicotinic skin reaction, also known as nicotinic flush reaction, occurs when a solution of nicotinic acid methyl ester briefly contacts the skin. Following penetration through the skin barrier into the subcutaneous tissue, it generates nicotinic acid (vitamin B3). Under the action of phospholipase A2 (PLA2), cyclooxygenase (COX), and other enzymes, arachidonic acid (AA) on the cell membrane is cleaved to produce prostaglandins, leading to local vasodilation, increased blood perfusion, and the transient appearance of erythema on the skin.

SUMMARY:
This study will explore the specific response characteristics of the niacin skin response test in the population with depressive disorder malinger. The investigators expect that depressive disorder malinger can be discriminated by the niacin skin reaction test.

DETAILED DESCRIPTION:
Depressive disorder malingers are prevalent, and it is difficult to recognize. As an objective and scientific endophenotype of depressive disorders, the blunted features in NSRT are determined by genetic factors and are not influenced by the mental state of individual subjects at a particular moment, which can provide a reliable retrospective biological index for the determination of mental and psychological state of depressive disorder malinger.

This study will explore the specific response characteristics of the niacin skin response test in the population with depressive disorder malinger, explore the application prospects of this technology in the field of biological identification, and establish a high-specificity biological diagnostic model for depressive disorder malinger and validate and optimize it, so as to provide a biological basis for the accurate and efficient identification of depressive disorder malingers using objective indexes in the process of clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Depressive Disorder Malinger Group:

1. Clinical complaints meeting DSM-5 criteria for the diagnosis of depressive disorder;
2. Patients with first-episode fraudulent disease who meet the DSM-5 criteria for the diagnosis of Z76.5;
3. Age 18-60 years, Males;
4. Voluntary informed consent.

Depressive Disorder Group:

1. Patients with a first depressive disorder meeting DSM-5 criteria;
2. Age 18-60 years, Males;
3. Voluntary informed consent.

Healthy control group:

1. M.I.N.I scale rating without any mental disorder;
2. PHQ-9 <5 ;
3. No history of mental illness, no family genetic history;
4. Age 18-60 years old, Males;
5. Voluntary informed consent form.

Exclusion Criteria:

1. History of traumatic brain injury;
2. Continuous use of non-steroidal anti-inflammatory drugs within the last two weeks.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Depressive Disorder Malinger Group
  2. Depressive Disorder Group
  3. Healthy Control Group
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Niacin reaction test | During the intervention
  Total niacin reaction score: It includes one value (Total Area), which refers to the sum of nicotinic acid reaction areas for each concentration (a total of 360) collected within 10 minutes from 60 images.
  Total single point score for niacin reaction: It includes six values, each representing the sum of nicotinic acid reaction areas for individual concentrations (a total of 360) collected within 10 minutes from 60 images.
  Niacin reaction speed: It includes one value (EC50), representing the time required for the nicotinic acid reaction of the first concentration to reach half of the plateau phase.
  Niacin flush color: It includes one value (Total Color), which refers to the color value of 6 flush areas in the images captured at the 10th minute.

SECONDARY OUTCOMES:
Model specificity and sensitivity | Through study completion, an average of 2 years
  Evaluate the effectiveness of the classification model in identifying feigned depression patients through measures such as the area under curve (AUC), sensitivity (Sen), specificity (Sep), positive predictive value (PPV), and negative predictive value (NPV), where higher AUC, Sen, Sep, PPV, and NPV values indicate better classification performance of the model.
The F Scale in Minnesota Multiphasic Personality Inventory | Baseline, pre-intervention
  The F Scale in Minnesota Multiphasic Personality Inventory (MMPI) is used to detect attempts at fraud.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Wang, Phd, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Air Force Medical Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated during and/or analysed during the current study will be available upon request from Jin Wang, sciaking@yeah.net

REFERENCES:
- [Background] Wang DD, Hu XW, Jiang J, Sun LY, Qing Y, Yang XH, Gao Y, Cui GP, Li MH, Wang PK, Zhang J, Zhuang Y, Li ZZ, Li J, Guan LL, Zhang TH, Wang JJ, Ji F, Wan CL. Attenuated and delayed niacin skin flushing in schizophrenia and affective disorders: A potential clinical auxiliary diagnostic marker. Schizophr Res. 2021 Apr;230:53-60. doi: 10.1016/j.schres.2021.02.009. Epub 2021 Mar 4. PMID 33677199
- [Background] Ward PE, Sutherland J, Glen EM, Glen AI. Niacin skin flush in schizophrenia: a preliminary report. Schizophr Res. 1998 Feb 9;29(3):269-74. doi: 10.1016/s0920-9964(97)00100-x. PMID 9516668
- [Background] Sun L, Yang X, Jiang J, Hu X, Qing Y, Wang D, Yang T, Yang C, Zhang J, Yang P, Wang P, Cai C, Wang J, He L, Wan C. Identification of the Niacin-Blunted Subgroup of Schizophrenia Patients from Mood Disorders and Healthy Individuals in Chinese Population. Schizophr Bull. 2018 Jun 6;44(4):896-907. doi: 10.1093/schbul/sbx150. PMID 29077970
- [Background] Messamore E, Hoffman WF, Yao JK. Niacin sensitivity and the arachidonic acid pathway in schizophrenia. Schizophr Res. 2010 Sep;122(1-3):248-56. doi: 10.1016/j.schres.2010.03.025. Epub 2010 Apr 24. PMID 20417059
- [Result] Wang J, Qing Y, Liang J, Cui G, Wang Q, Zhang J, Yang X, Li M, Wang D, Fan Z, Chu K, Zhang J, Ke X, Wan C. Identification of adolescent patients with depression via assessment of the niacin skin flushing response. J Affect Disord. 2023 Mar 1;324:69-76. doi: 10.1016/j.jad.2022.12.017. Epub 2022 Dec 12. PMID 36521667